CLINICAL TRIAL: NCT00237354
Title: A Phase 1 Safety and Tolerability Study of PV-10 Chemoablation of Recurrent Breast Carcinoma
Brief Title: PV-10 Chemoablation of Recurrent Breast Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Provectus Pharmaceuticals (Industry)
Responsible Party: Eric Wachter, Ph.D., Provectus Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PV-10-BC-04
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Breast Cancer
Keywords: Recurrent soft tissue breast carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Rose Bengal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PV-10 (rose bengal disodium 10%) — PV-10 ablation of study lesion

SUMMARY:
The objective of this study is to investigate the safety of intralesional (IL) PV-10 for the treatment of recurrent breast carcinoma. This study will also include a preliminary assessment of response of injected lesions by histologic assessment upon lesion excision at 1-3 weeks following IL PV-10 administration. Post-excision wound healing will be assessed clinically at 1 week and 4 weeks following excision of PV-10 injected lesions.

DETAILED DESCRIPTION:
This is a single center, open label, ascending dose study. Subjects with at least one recurrent, histologically confirmed measurable soft tissue breast carcinoma who are candidates for lumpectomy (removal of the lesion from the site of recurrence in the breast or at another site) or mastectomy will receive a single intralesional injection of PV-10 into a single target lesion to uniformly infiltrate the target lesion and up to a 0.5 cm margin at a dose of up to 1.0 mL/cc lesion volume. Systemic and locoregional adverse events will be monitored over the study interval. Subject accrual and PV-10 administration will be stopped if more than 1 subject has a treatment related Grade 3 non-hematological or Grade 4 hematological toxicity within a period of two weeks after PV-10 administration.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed recurrent soft tissue breast carcinoma
* At least one measurable target lesion at least 0.5 cm and no more than 3 cm in longest diameter
* Performance Status: Karnofsky 70-100% or ECOG 0-2
* Life Expectancy: At least 6 months
* Hematopoietic:

  * White blood cell count (WBC) at least 3000/mm3
  * Absolute neutrophil count (ANC) at least 1.5 (1,500/mm3)
  * Hemoglobin at least 10 g/dL
  * Platelet count at least 100,000/mm3
* Coagulopathy: International Normalized Ratio (INR) at least 1.5.
* Renal Function: Creatinine = 0.05-0.11 mmol/L
* Hepatic Function:

  * Bilirubin = 3-21 umol/L
  * AST/ALT ≤ 3 times the upper limit of normal (ULN)
* Cardiovascular Function: No major cardiovascular disease
* Thyroid Function: T3 (serum triiodothyronine), T4 (serum thyroxine) and THS (serum thyrotropin) within normal limits
* Immunological Function: Adequate immune system function in the opinion of the investigator

Exclusion Criteria:

* Radiation therapy to study lesions within 4 weeks
* Chemotherapy or other systemic cancer therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin)
* Local treatment (e.g., surgery, cryotherapy, radiofrequency ablation) to the treatment area within 4 weeks
* Investigational agents within 4 weeks (or 5 half-lives)
* Anti-tumor vaccine therapy within 12 weeks
* Concurrent illness:

  * Severe diabetes or extremity complications due to diabetes
  * Significant concurrent disease or illness, psychiatric disorders, or alcohol or chemical dependence that would, in the opinion of the investigator, compromise subject safety or compliance or interfere with interpretation of study results
  * Thyroid autoregulatory dysfunction, including thyroid disease (subclinical or ongoing), goiter, partial thyroidectomy, prior radioiodine- or surgically-treated Graves' hyperthyroidism, or cystic fibrosis
* Pregnancy or fertile female subjects who are not using effective contraception, or who are lactating
* Known or suspected brain metastases or spinal cord compression.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Systemic and locoregional adverse experience | 5-7 weeks post dosing (4 weeks post excision)

SECONDARY OUTCOMES:
Histopathologic response of PV-10 injected lesions | 7-21 days post dosing
Wound healing of PV-10 injected lesions | 5-7 weeks post dosing (4 weeks post excision)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wachter, Ph.D., Study Director — Provectus Pharmaceuticals, Inc.; Chris Wynne, M.D., Principal Investigator — Oncology Service, Christchurch Hospital
Locations (1):
- Canterbury BreastCare, Christchurch, New Zealand